CLINICAL TRIAL: NCT06261372
Title: The Influence of Mindfulness Meditation Combined With Progressive Muscle Relaxation Training on the Clinical Efficacy and Quality of Life of Hemodialysis Patients With Sarcopenia
Brief Title: Mindfulness Meditation Combined With Progressive Muscle Relaxation Training for Uremic Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2023PJ204
Record Dates: First submitted 2024-01-13; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Hemodialysis Patients With Sarcopenia
Keywords: mindfulness meditation; progressive muscle relaxation; uremic sarcopenia; maintenance hemodialysis; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group received conventional dialysis treatment.
- intervention group (Other): In addition to conventional treatment, mindfulness meditation combined with progressive muscle relaxation training was implemented during the interdialytic period.
  Interventions: Behavioral: The mindfulness meditation combined with progressive muscle relaxation training .

INTERVENTIONS:
Behavioral: The mindfulness meditation combined with progressive muscle relaxation training . — The first part is progressive muscle relaxation training. The second part is mindfulness meditation training.
  Arms: intervention group

SUMMARY:
To study the effect of mindfulness meditation combined with progressive muscle relaxation training on clinical efficacy and quality of life in maintenance hemodialysis (MHD) patients with sarcopenia. Eligible sarcopenic patients in our hospital were randomly assigned to a control group (n = 24) and an intervention group (n = 25). The control group received conventional dialysis treatment, while the intervention group received mindfulness meditation combined with progressive muscle relaxation training during the interdialysis period in addition to conventional dialysis treatment. The effect of the intervention was evaluated after 12 weeks.To observe whether the combined intervention training can improve the motor ability and quality of life of patients with sarcopenia in a short period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the sarcopenia criteria established by the Asian Working Group for Sarcopenia (AWGS) in 2014
* Stable condition and generally good health status
* Good compliance and ability to collaborate well with the physician
* Undergoing hemodialysis three times per week for at least three months, with a KT/V ≥ 1.2
* No significant cardiovascular or cerebrovascular complications (such as severe heart failure, severe arrhythmias, angina, and cerebrovascular diseases)
* Patients with sarcopenia who met the clinical diagnostic criteria were selected to ensure the quality of the included patients

Exclusion Criteria:

* Inability to complete handgrip strength, 6-meter walk test, 10 sit-to-stand tests, and the use of bioelectrical impedance analysis (BIA) due to contraindications
* Coexistence of mental illness or severe cognitive or communication disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
10 sit-to-stand test in seconds | 3 months
  The 10 sit-stand test represents exercise ability, and the shorter the time, the greater the exercise ability.
Grip strength in kilograms | 3 months
  Grip strength represents exercise ability, and the larger it is, the more exercise ability it is.Its minimum value is zero, and its maximum value is unlimited.
6-meter walk test in metre per second | 3 months
  6-meter walk test represents exercise ability, and the larger it is, the more exercise ability it is.Its minimum value is zero metre per second, and its maximum value is unlimited.
KDQOLTM(Kidney Disease Quality of Life short Form) score | 3 months
  The KDQOLTM score is between 0 and 100, and the higher the score, the better the health
interleukin-6 (IL-6) | 3 months
  Interleukin 6 represents an inflammatory marker, and its concentration is 20pg/ml or less.
high-sensitivity C-reactive protein (hsCRP) | 3 months
  hsCRP represents an inflammatory marker, and its concentration ranges from 0.0 to 10mg/L.
albumin(ALB) | 3 months
  Albumin represents a nutritional indicator, and its concentration ranges from 40 to 55g/L.
prealbumin (PA） | 3 months
  Prealbumin represents a nutritional indicator, and its concentration ranges from 0.20 to 0.43g/l.

CONTACTS AND LOCATIONS:
Locations (1):
- Li Huili Hospital, Ningbo Medical Center, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Y, Zhang H, Jiang L, Liu Z, Li X, Guo B, Li J, Xu P, Liu J, Yu R. Effects of mindfulness meditation combined with progressive muscle relaxation on sleep disorders, anxiety, and depression in patients with sarcopenia undergoing hemodialysis. Front Psychiatry. 2025 Jun 13;16:1542028. doi: 10.3389/fpsyt.2025.1542028. eCollection 2025. PMID 40585548